CLINICAL TRIAL: NCT00131911
Title: A Phase II Trial of Bay 43-9006 in Progressive Metastatic Neuroendocrine Tumors
Brief Title: Sorafenib Tosylate in Treating Patients With Progressive Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00121; MC044H; 7046; CDR0000437792; N01CM62205 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-06

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Metastatic Gastrointestinal Carcinoid Tumor; Neuroendocrine Tumor; Pancreatic Polypeptide Tumor; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma; Somatostatinoma; WDHA Syndrome
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Neuroendocrine Tumors; Carcinoma, Islet Cell; Somatostatinoma; Vipoma | interventions — Sorafenib

ARMS (2):
- Group A (patients with carcinoid tumors) (Experimental): Patients receive 400 mg oral sorafenib twice daily on days 1-28.
  Interventions: Drug: sorafenib tosylate
- Group B (islet cell and other neuroendocrine tumors) (Experimental): Patients receive 400 mg oral sorafenib twice daily on days 1-28.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — 400 mg given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
This phase II trial is studying how well sorafenib tosylate works in treating patients with progressive metastatic neuroendocrine tumors. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective tumor response rate of BAY 43-9006 (sorafenib tosylate) in patients with advanced neuroendocrine tumors.

SECONDARY OBJECTIVES:

I. Adverse event rate(s). II. Progression free survival and time to progression. III. Improvement in circulating hormone levels. IV. Overall survival.

OUTLINE: This is a multicenter study. Patients are grouped into 2 separate analysis Groups according to tumor type (Group A: Carcinoid; Group B: Islet cell/other well-differentiated tumor). Each Group was independently evaluated for all study endpoints.

Patients receive oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 2 years from study entry.

ELIGIBILITY:
Criteria:

* Histologically confirmed neuroendocrine tumor:

  * Carcinoid tumor OR islet cell carcinoma/other well-differentiated tumor
  * No anaplastic or high-grade histology
  * Metastatic disease
* Measurable disease
* No thyroid carcinoma of any histology, thymoma, or pheochromocytoma/paraganglioma
* No known brain metastases
* Performance status:

  * Eastern Cooperative Oncology Group (ECOG) 0-2
* Life expectancy:

  * At least 24 weeks
* Hematopoietic:

  * Absolute neutrophil count >= 1,500/mm3
  * Platelet count >= 100,000/mm3
  * No bleeding diathesis
* Hepatic:

  * Bilirubin =< 2 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) =< 3 times ULN (5 times ULN if liver metastases are present)
  * International normalized ratio (INR) normal
  * PTT normal
* Renal:

  * Creatinine =< 1.5 times ULN
* Cardiovascular:

No poorly controlled hypertension; No symptoms of congestive heart failure; No unstable angina pectoris; No cardiac arrhythmia

* Gastrointestinal:

  * Able to swallow capsules intact
  * No gastrointestinal tract disease resulting in an inability to take oral medication (e.g., dysphagia)
  * No requirement for IV alimentation
  * No active peptic ulcer disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other invasive malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other uncontrolled illness
* At least 4 weeks since prior interferon
* No more than 1 prior systemic chemotherapy regimen:

Chemoembolization is not considered systemic chemotherapy

* At least 4 weeks since prior chemoembolization
* At least 3 weeks since prior radiotherapy
* No prior procedures adversely affecting intestinal absorption
* At least 4 weeks since prior hepatic artery embolization
* No other prior systemic therapy
* No other concurrent investigational treatment
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent enzyme-inducing anticonvulsants (e.g., carbamazepine, phenobarbital, or phenytoin)
* No concurrent rifampin
* No concurrent Hypericum perforatum (St. John's wort)
* Prior or concurrent octreotide for symptomatic treatment allowed
* No concurrent therapeutic anticoagulation:

Concurrent prophylactic anticoagulation (i.e., low dose warfarin) of venous or arterial access devices allowed provided requirements for INR or PTT are met

* At least 4 weeks since prior major surgery
* Recovered from all prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2005-06; Primary Completion 2010-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Hobday, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 21, 2005 and September 15, 2006, a total of 93 (51 carcinoid, 42 islet cell) patients initiated treatment on this study.
Pre-assignment Details: One carcinoid patient canceled prior to treatment and was excluded from all analyses.
Period: Overall Study
Arm/Group | Group A (Patients With Carcinoid Tumors) | Group B (Islet Cell and Other Neuroendocrine Tumors)
Started | 51 | 42
Completed | 50 | 42
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Patients With Carcinoid Tumors) | Group B (Islet Cell and Other Neuroendocrine Tumors) | Total
Number analyzed (Participants) | 51 | 42 | 93
Age, Continuous [Median (Full Range); unit: years] | 60 [38 to 82] | 56.5 [26 to 78] | 59 [26 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 49
  Male | 23 | 21 | 44
Region of Enrollment [Number; unit: participants]
  United States | 51 | 42 | 93

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate
Description: Confirmed response rate was defined using Response Evaluation Criteria In Solid Tumors (RECIST). A confirmed response is defined as a complete response (CR) or partial response (PR) observed on subsequent scans at least 4 weeks apart. Confirmed response rate was estimated by the number of successes divided by the total number of evaluable patients.> > Complete Response (CR) is defined as the disappearance of all target lesions.> Partial Response (PR) is defined as a 30% decrease in sum of longest diameter of target lesions;>
  > We report the percentage of patients with a confirmed response and a 95% confidence interval estimated by the Duffy and Santner method.
Time Frame: Duration of Treatment (Up to 2 years)
Population: Nine of the 50 carcinoid patients and 6 of the 42 Islet cell patients did not continue treatment past cycle 1. Therefore, these patients were not evaluated on consecutive cycles and were excluded from this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Patients With Carcinoid Tumors) | Group B (Islet Cell and Other Neuroendocrine Tumors)
Number analyzed (Participants) | 41 | 36
percentage of participants | 10 [3 to 24] | 14 [6 to 32]

2. Secondary Outcome: Toxicity
Description: For this secondary endpoint, toxicity is defined as a grade 3 or higher adverse events that is classified as either possibly, probably, or definitely related to study treatment. The assignment of attribution to study treatment and grade (or degree of severity) of the adverse event are classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The number of participants reporting a grade 3 or higher toxicity are reported.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Group A (Patients With Carcinoid Tumors) | Group B (Islet Cell and Other Neuroendocrine Tumors)
Number analyzed (Participants) | 50 | 42
participants
  Grade 3 Toxicity | 37 | 25
  Grade 4 or Grade 5 Toxicity | 5 | 2

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from registration to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: From registration to death (up to 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A (Patients With Carcinoid Tumors) | Group B (Islet Cell and Other Neuroendocrine Tumors)
Number analyzed (Participants) | 50 | 42
months | 25.6 [15.5 to 30.2] | NA [NA to NA] — At the time of analysis, a sufficient number of events had not been recorded to estimate.

4. Secondary Outcome: Progression Free Survival
Description: Progression was defined using Response Evaluation Criteria In Solid Tumors (RECIST) as a 20% increase in the su of longest diameter of target lesions. Progression free survival (PFS) was defined as the time from registration to progression or death of any cause. Participants who were progression free were censored at the date of their most recent disease assessment. The median PFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Time from registration to progression or death (up to 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A (Patients With Carcinoid Tumors) | Group B (Islet Cell and Other Neuroendocrine Tumors)
Number analyzed (Participants) | 50 | 42
months | 9.1 [5.7 to 12.7] | 12.7 [8.3 to 19.9]

5. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the time from attaining a response (PR or CR) to the date of progression. Participants without progression were censored at the date of their most recent disease assessment. The median DOR was estimated using simple summary statistics.
Time Frame: Time from response to progression (up to 2 years)
Population: There were 4 confirmed responses in Group A and 5 confirmed responses in Group B used in analyzing this endpoint.
Measure: Median (Full Range); unit: months
Arm/Group | Group A (Patients With Carcinoid Tumors) | Group B (Islet Cell and Other Neuroendocrine Tumors)
Number analyzed (Participants) | 4 | 5
months | 6.7 [3.7 to 9.2] | 9.2 [3.7 to 32]

ADVERSE EVENTS:
Groups:
- All Patients: Patients receive 400 mg oral sorafenib twice daily on days 1-28.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 52/93
Other Adverse Events (participants affected / at risk) | 90/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=93)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 18 (22)
Ascites (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 13 (15)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (5)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 15 (15)
Fever (General disorders) | 4 (4)
Localized edema (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (3)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 10 (11)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 6 (7)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (6)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3)
Flushing (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=93)
Blood disorder (Blood and lymphatic system disorders) | 2 (7)
Hemoglobin decreased (Blood and lymphatic system disorders) | 18 (63)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Hearing test abnormal (Ear and labyrinth disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 1 (37)
Diplopia (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (2)
Retinal detachment (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 5 (16)
Abdominal pain (Gastrointestinal disorders) | 34 (99)
Anal pain (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 65 (467)
Dry mouth (Gastrointestinal disorders) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 10 (40)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 35 (99)
Flatulence (Gastrointestinal disorders) | 9 (88)
Gingival pain (Gastrointestinal disorders) | 1 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 45 (121)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (5)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (31)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 5 (8)
Edema limbs (General disorders) | 8 (10)
Fatigue (General disorders) | 63 (306)
Fever (General disorders) | 8 (10)
Localized edema (General disorders) | 3 (3)
Pain (General disorders) | 4 (27)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 4 (7)
Anal infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Prostate infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 4 (16)
Upper respiratory infection (Infections and infestations) | 4 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 21 (88)
Alkaline phosphatase increased (Investigations) | 28 (163)
Aspartate aminotransferase increased (Investigations) | 32 (115)
Blood bilirubin increased (Investigations) | 7 (14)
Blood corticotrophin decreased (Investigations) | 1 (1)
Creatine phosphokinase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 14 (33)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 2 (6)
Leukocyte count decreased (Investigations) | 8 (11)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (12)
Neutrophil count decreased (Investigations) | 5 (8)
Platelet count decreased (Investigations) | 24 (67)
Serum cholesterol increased (Investigations) | 1 (1)
Weight loss (Investigations) | 10 (27)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 39 (100)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 7 (13)
Blood glucose increased (Metabolism and nutrition disorders) | 11 (31)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (45)
Serum calcium decreased (Metabolism and nutrition disorders) | 11 (23)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 5 (8)
Serum phosphate decreased (Metabolism and nutrition disorders) | 6 (9)
Serum potassium decreased (Metabolism and nutrition disorders) | 6 (8)
Serum potassium increased (Metabolism and nutrition disorders) | 5 (9)
Serum sodium decreased (Metabolism and nutrition disorders) | 7 (9)
Serum sodium increased (Metabolism and nutrition disorders) | 5 (9)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (17)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (64)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Accessory nerve disorder (Nervous system disorders) | 1 (10)
Dizziness (Nervous system disorders) | 6 (16)
Dysgeusia (Nervous system disorders) | 3 (11)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (16)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (8)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (14)
Confusion (Psychiatric disorders) | 1 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (11)
Hemoglobin urine positive (Renal and urinary disorders) | 3 (4)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 (73)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 (27)
Alopecia (Skin and subcutaneous tissue disorders) | 46 (246)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (29)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 52 (267)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (5)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 51 (184)
Rash desquamating (Skin and subcutaneous tissue disorders) | 15 (21)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Sweating (Skin and subcutaneous tissue disorders) | 6 (11)
Flushing (Vascular disorders) | 6 (15)
Hot flashes (Vascular disorders) | 6 (12)
Hypertension (Vascular disorders) | 51 (189)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less